CLINICAL TRIAL: NCT03292094
Title: African Prospective Study for the Early Detection and Identification of Cardiovascular Disease and Hypertension (African-PREDICT Study)
Brief Title: The African-PREDICT Study
Acronym: PREDICT
Status: Active, not recruiting | Type: Observational
Sponsor: North-West University, South Africa (Other)
Collaborators: Medical Research Council, South Africa (Other); National Research Foundation of South Africa (Other); GlaxoSmithKline (Industry); Medical Research Council (Other Government); Pfizer (Industry); Boehringer Ingelheim (Industry); Novartis (Industry); Mediclinic Hospital (Unknown); Roche Diagnostics GmbH (Industry)
Responsible Party: Principal Investigator, Alta Schutte, Professor, North-West University, South Africa
Other Study IDs: NWU-00001-12-A1
Record Dates: First submitted 2017-09-12; First posted 2017-09-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Cardiovascular Diseases; Hypertension; Health Risk Behaviors; Arterial Stiffness; Young; Renin Hypertension
Keywords: Young; Healthy; African; Longitudinal; Hypertension; Salt intake; Obesity; Organ damage
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Health Risk Behaviors; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological samples for biomarker analyses (serum, plasma, spot urine and 24-hr urine) were taken at baseline and each follow-up. Samples are preserved for the short and long-term at -80°C. We will assess a wide range of traditional and novel biomarkers related to hypertension and cardiovascular disease. These samples will also be analysed in an attempt to identify bio-signatures in terms of the -omics sciences (genomic, metabolomic and proteomic profiles) as predictors of cardiovascular deterioration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Black men: 294 young healthy men were included (clinic normotensive, non-HIV)
- White men: 284 young healthy men were included (clinic normotensive, non-HIV)
- Black women: 312 young healthy women were included (clinic normotensive, non-HIV)
- White women: 312 young healthy women were included (clinic normotensive, non-HIV)

SUMMARY:
The African-PREDICT study aims to (i) generate new knowledge on the early pathophysiology accompanying hypertension development in black South Africans; and (ii) to identify early novel markers or predictors for the development of hypertension and cardiovascular outcome. By employing also in Africa the latest cutting-edge scientific technologies to measure single and multiple biomarkers proven to predict hypertension and cardiovascular outcome (such as multiplex analyses, proteomics and metabolomics), precision medicine may have the potential to lead to novel strategies in preventing and treating hypertension in Africa.

DETAILED DESCRIPTION:
Background and Problem Statement: Recent global analyses have indicated that the highest blood pressures worldwide are recorded in black populations. The vulnerable cardiovascular profile of Africans is believed to result from a combination of factors such as rapid urbanisation, abnormal sodium handling, elevated vascular resistance and arterial stiffness. The frequent underdiagnoses and ineffective treatment of hypertension in general but especially in Africans, result in severe complications, such as stroke, heart and kidney disease. Since diagnosis and treatment are generally unsuccessful in black populations - especially in low and middle-income countries - prevention is key to curb the rapidly increasing incidence of death and disability from cardiovascular disease. Cardiovascular risk prediction in black populations worldwide is inadequate since we do not have a clear understanding of the complex mechanisms underlying the development of cardiovascular disease.

Main Aim: In the "African PRospective study on the Early Detection and Identification of Cardiovascular disease and Hypertension" (African-PREDICT) the investigators aim to identify early markers or predictors for the development of cardiovascular disease in black South Africans. Only by understanding the early pathophysiology of disease development, and by identifying markers as potential screening indicators, predictors or targets for intervention, will the investigators be able to implement successful prevention programes in Africans at younger ages. The researchers therefore aim to track and monitor change in young, normotensive black and white individuals (aged 20-30 years) over 10-20 years. To achieve this the investigators will perform detailed cardiovascular and novel biomarker measurements, as well as behavioural and biopsychosocial assessments every 4-5 years in order to identify and understand early changes in cardiovascular function, and specific predictors contributing to the development of hypertension and target organ damage.

Methodology and Measurements: In 2013 recruitment started, screening and assessment of 1200 normotensive and apparently healthy participants (black N=600 and white N=600) with equal sex distribution. A wide range of basic and advanced measurements are taken within a Hypertension Clinic to get a highly detailed profile of the participants at each visit. The following is obtained: (1) relevant questionnaire data including medical history, lifestyle, social status, traditional risk factors (age, gender, smoking, alcohol intake) and validated questionnaires on dietary intake, personality and psychosocial profile; (2) Biological samples for biomarker analyses (serum, plasma, spot urine and 24-hr urine) are taken and preserved for the short and long-term at -80°C. A wide range of traditional and novel biomarkers related to hypertension and cardiovascular disease (including amongst others, lipid profile, glucose, glycated hemoglobin, C-reactive protein, interleukin-6, vitamin D, full blood count, sodium, potassium, creatinine, renin, aldosterone, angiotensin II, markers of oxidative stress and nitric oxide bio-availability, cortisol, sex hormones, insulin, C-peptide, leptin and other adipokines, angiogenic markers, the insulin-like growth factor-axis, soluble urokinase plasminogen activator receptor, Nt-proBNP, fibulin-1 and novel markers not yet identified) will be assessed. These samples will also be analysed in an attempt to identify bio-signatures in terms of the -omics sciences (genomic, metabolomic and proteomic profiles) as predictors of cardiovascular deterioration; (3) anthropometric measurements, bio-electrical impedance measurement of body fat and lean mass, and 7-day physical activitymonitoring; (4) A range of cardiovascular assessments: 24-hour blood pressure, central arterial pressure, and cardiovascular stress reactivity tests with continuous finger blood pressure; and (5) Assessments of early target organ damage including urinary albumin-to-creatinine ratio, carotid intima-media thickness, ECG, echocardiography, pulse wave velocity, and retinal microvascular calibre and dilation during provocation with a light flicker test.

Timetable: The project was approved and is endorsed by the National and Provincial Department of Health, and was approved by the Ethics Committee of the North-West University in 2012 (NWU-00001-12-A1). Screening commenced in November 2012, and research participants started entering the study from 6 February 2013. Baseline data collection was completed in December 2017. Follow-up assessments commenced in February 2018 and will continue until Dec 2022. The Health Research Ethics Committee approved continuation of the study for 2020.

Anticipated Outcomes: This project will increase understanding of the complex mechanisms involved in the aetiology of early cardiovascular changes in relatively young individuals from African and European ancestry, which will (1) improve ability to identify individuals at risk before the development of cardiovascular diseases (CVD), and (2) predict the development of future hypertension and related CVD. Both outcomes will make it possible to develop better individualised and population-based prevention of CVD contributing to better quality of life. These results will not only be applicable to Sub-Saharan Africa but are expected to have a broader impact with regards to white and black populations globally. Results are expected to have significant scientific impact by means of publications in high-impact journals; and also to translate directly into novel preventive healthcare policy and practices - translating into preventive measures regarding the development of CVDs in clinics throughout South Africa.

ELIGIBILITY:
Inclusion Criteria:

* Brachial BP <140 and 90 mmHg
* HIV uninfected
* No previous diagnosis or medication for chronic disease
* Not pregnant or breastfeeding

Exclusion Criteria:

* Planning to move away from the Potchefstroom area in the next 5 years
* Currently pregnant or breastfeeding
* Sick on the day of appointment
* Lack the ability to read or understand English
* Diagnosed with HIV, Cancer, Tuberculosis, Diabetes, Hypertension, Liver or Kidney disease, Heart disease
* Previously had a heart attack or stroke
* Have suffered a recent trauma or had surgery in the past 3 months
* Have a phobia for needles
* Have donated blood in the previous 3 months
* Taking chronic medication (Anti-inflammatory, for Hypertension of Diabetes, Cortisone, Anti-Retroviral, Thyroid medication, Cholesterol medication)

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Apparently healthy black and white participants between the ages of 20 and 30 years from the Potchefstroom area, North West Province, South Africa.
Sampling Method: Non-Probability Sample
Enrollment: 1202 (Actual)
Dates: Start 2013-02-04 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2027-12-03 (Estimated)

PRIMARY OUTCOMES:
Incident Hypertension | 5 years
  Incident hypertension based on 4 repeated clinic blood pressure measurements, i.e. SBP>=140 mmHg and/or DBP >=90 mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Alta Schutte, PhD, Principal Investigator — University of New South Wales; Carina MC Mels, PhD, Principal Investigator — North-West University
Locations (1):
- Hypertension Research and Training Clinic, Potchefstroom, North West, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mokgonyana PJ, Mokwatsi GG, Gwini SM, Gafane-Matemane LF. The relationship between kidney function and the soluble (pro)renin receptor in young adults: the African-PREDICT study. BMC Nephrol. 2025 Apr 3;26(1):172. doi: 10.1186/s12882-025-04038-x. PMID 40181300
- [Derived] Degenaar A, Kruger R, Jacobs A, Mels CMC. Phenotyping Kidney Function in Young Adults With High Blood Pressure: The African-PREDICT Study. J Clin Hypertens (Greenwich). 2024 Nov;26(11):1291-1300. doi: 10.1111/jch.14911. Epub 2024 Oct 5. PMID 39368068
- [Derived] Strauss-Kruger M, Pieters M, van Zyl T, Gafane-Matemane LF, Mokwatsi GG, Jacobs A, Schutte AE, Louw R, Mels CM. Metabolomic Insights on Potassium Excretion, Blood Pressure, and Glucose Homeostasis: The African-PREDICT Study. J Nutr. 2024 Feb;154(2):435-445. doi: 10.1016/j.tjnut.2023.12.025. Epub 2023 Dec 16. PMID 38110181
- [Derived] Gafane-Matemane LF, Kruger R, Smith W, Mels CMC, Van Rooyen JM, Mokwatsi GG, Uys AS, Brits SJ, Schutte AE. Characterization of the Renin-Angiotensin-Aldosterone System in Young Healthy Black Adults: The African Prospective Study on the Early Detection and Identification of Hypertension and Cardiovascular Disease (African-PREDICT Study). Hypertension. 2021 Aug;78(2):400-410. doi: 10.1161/HYPERTENSIONAHA.120.16879. Epub 2021 Jun 28. PMID 34176281
- [Derived] Kochli S, Schutte AE, Botha-Le Roux S, Gafane-Matemane LF, Smith W, van Rooyen JM, Mokwatsi GG, Kruger R. Potassium excretion and blood pressure are associated with heart rate variability in healthy black adults: The African-PREDICT study. Nutr Metab Cardiovasc Dis. 2021 Apr 9;31(4):1071-1080. doi: 10.1016/j.numecd.2020.12.021. Epub 2020 Dec 24. PMID 33549447
- [Derived] Crouch SH, Botha-Le Roux S, Delles C, Graham LA, Schutte AE. Inflammation and hypertension development: A longitudinal analysis of the African-PREDICT study. Int J Cardiol Hypertens. 2020 Dec;7:100067. doi: 10.1016/j.ijchy.2020.100067. PMID 33392493

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/94/NCT03292094/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/94/NCT03292094/ICF_001.pdf